CLINICAL TRIAL: NCT05175898
Title: Treatment With Leftventricular Impella® Micro-axial Pump and Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO) During Extracorporeal Cardiopulmonary Resuscitation (eCPR) on Mortality - An International Multicenter Cohort Study
Brief Title: ECMELLA vs. ECMO on 30-day Mortality
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Carsten Skurk, Professor, Charite University, Berlin, Germany
Other Study IDs: ECMELLA vs. ECMO
Record Dates: First submitted 2021-10-27; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest; Extracorporeal Membrane Oxygenation Complication; Cardiogenic Shock; Acute Myocardial Infarction
MeSH Terms: conditions — Heart Arrest; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VA-ECMO: Patients who were treated with veno-arterial extracorporeal membrane oxygenation (VA-ECMO) during cardiac arrest.
  Interventions: Device: VA-ECMO
- ECMELLA: Patients who were treated with veno-arterial extracorporeal membrane oxygenation (VA-ECMO) and Impella® micro-axial pump.
  Interventions: Device: ECMELLA

INTERVENTIONS:
Device: VA-ECMO — Treatment with veno-arterial extracorporeal membrane oxygenation
  Groups: VA-ECMO
Device: ECMELLA — Treatment with veno-arterial extracorporeal membrane oxygenation plus Impella® micro-axial pump.
  Groups: ECMELLA

SUMMARY:
This international, multicenter cohort study aims to investigate outcomes after treatment with extracorporeal cardiopulmonary resuscitation (eCPR) during cardiac arrest.

DETAILED DESCRIPTION:
Left ventricular unloading with Impella® micro-axial pump has been shown to improve survival in patients with cardiogenic shock treated with veno-arterial extracorporeal membrane oxygenation (VA-ECMO). This study aims to investigate whether treatment with VA-ECMO and Impella ® (so called "ECMELLA") during extracorporeal cardiopulmonary resuscitation is associated with improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Cardiac arrest
* Treatment with veno-arterial extracorporeal membrane oxygenation (VA-ECMO) or "ECMELLA" (that is VA-ECMO plus left ventricular Impella® micro-axial pump)

Exclusion Criteria:

* Non-adult patients
* No treatment with VA-ECMO or "ECMELLA"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were treated with veno-arterial extracorporeal membrane oxygenation (VA-ECMO) or VA-ECMO and Impella (so called "ECMELLA") during extracorporeal cardiopulmonary resuscitation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | Mortality within 30 days after cardiac arrest event.
  Mortality within 30 days after cardiac arrest event.

SECONDARY OUTCOMES:
Hospital length of stay | Through study completion - an average of 1 year.
  Number of days between hospital admission and hospital discharge.
Intensive Care Unit (ICU) length of stay | Through study completion - an average of 1 year.
  Number of ICU days between ICU admission and ICU discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skurk, MD, Principal Investigator — Charite University; Tharusan Thevathasan, MD, Principal Investigator — Charite University
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No